CLINICAL TRIAL: NCT00623883
Title: Colonoscopic Biomarkers for Cancer Risk Assessment and Prevention
Brief Title: Colonoscopic Removal of Aberrant Crypt Foci: a Prospective, Randomized, Blinded Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Naval Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Peter W. Soballe, CAPT, MC, USN, National Naval Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NNMC.1997.0091
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2007-06

CONDITIONS: Colorectal Neoplasms
Keywords: Human Colonic Aberrant Crypt Foci
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): All identified ACF eliminated by cold or hot colonoscopic biopsy forceps
  Interventions: Procedure: Surgical removal of ACF
- 2 (Sham Comparator): ACF quantified and observed, re-evaluated after one year
  Interventions: Procedure: Colonoscopic evaluation only

INTERVENTIONS:
Procedure: Surgical removal of ACF — All ACF removed by either cold or hot colonoscopic biopsy forceps
  Arms: 1
Procedure: Colonoscopic evaluation only — Stain-enhanced magnification endoscopy performed, ACF quantified at entry and after one year
  Arms: 2

SUMMARY:
We hypothesized that aberrant crypt foci (ACF) are precursors of colon cancer; their prevention would correlate with cancer risk and their elimination would reduce that risk. In this study we wished to (1) establish the feasibility of stain-enhanced magnification colonoscopy, (2) determine whether colorectal cancer is asociated with increased numbers of ACF, and (3) investigate the natural history of ACF and the durability of their elimination.

DETAILED DESCRIPTION:
Subjects are randomly assigned at the time of stain-enhanced magnification colonoscopy to have any ACF removed or merely observed. Subjects are evenly divided into those with and those without a personal history of colon cancer. ACF are tabulated by an observer blinded to the subject's personal history. All subjects are then re-evaluated after one year by an observer blinded to the original procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Dept.of Defense Healthcare Beneficiaries
2. Age 18 or over, non-pregnant
3. History of colorectal cancer or other indication for colonoscopic screening
4. At least half of large intestine remaining
5. No use of investigational or chemotherapeutic drugs within 6 mos. -

Exclusion Criteria:

1. History suggesting familial colon cancer syndrome
2. < 6 mos since colon resection or since treatment for colon cancer
3. Anticipated colon surgery within one year of entry
4. Inability to participate in scheduled followup at one year
5. Medical or psychiatric condition which would make patient a poor candidate -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 1999-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
number, size, and location of ACF identified | initially and after one year

SECONDARY OUTCOMES:
complications of stain-enhanced, magnification colonoscopy | initially and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Soballe, M.D., Principal Investigator — National Naval Medical Center
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Result] Glebov OK, Rodriguez LM, Soballe P, DeNobile J, Cliatt J, Nakahara K, Kirsch IR. Gene expression patterns distinguish colonoscopically isolated human aberrant crypt foci from normal colonic mucosa. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2253-62. doi: 10.1158/1055-9965.EPI-05-0694. PMID 17119054
- [Result] Glebov OK, Rodriguez LM, Nakahara K, Jenkins J, Cliatt J, Humbyrd CJ, DeNobile J, Soballe P, Simon R, Wright G, Lynch P, Patterson S, Lynch H, Gallinger S, Buchbinder A, Gordon G, Hawk E, Kirsch IR. Distinguishing right from left colon by the pattern of gene expression. Cancer Epidemiol Biomarkers Prev. 2003 Aug;12(8):755-62. PMID 12917207